CLINICAL TRIAL: NCT02621437
Title: Study of the Impact of Osteopathic Care, Complementary Therapy to Standard Care, on Pain in Patients With Breast Cancer Surgery
Brief Title: Impact of Osteopathy on Pain After Breast Cancer Surgery
Acronym: IPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69HCL14_0456
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: pain; quality of life; osteopathy; oncology; surgery; breast
MeSH Terms: conditions — Breast Neoplasms; Pain; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (osteopathy) (Experimental): Patients will have three sessions of osteopathy and 6 phone questionnaires.
  Interventions: Other: Osteopathy sessions; Other: phone questionnaires
- control group (Other): Patients will have 6 phone questionnaires.
  Interventions: Other: phone questionnaires

INTERVENTIONS:
Other: Osteopathy sessions — - Three osteopathy sessions every 14 days (D13, D27 and D41 post-surgery),
  Arms: Intervention group (osteopathy)
Other: phone questionnaires — Six phone questionnaires (D9, D20, D26, D34, D40 and D48):
  * pain questionnaire with digital scale,
  * quality of life survey: SF-12
  * HAD (Hospital and Anxiety Depression) questionnaire

SUMMARY:
Breast cancer can be painful following surgery or can develop later and remain persistent. Pain occurrence is frequent with 50% of women developing sequelae pain of varying intensity with an impact on the quality of life. One of the priorities of the 3rd French Cancer Plan is to preserve quality of life.

Osteopathy, complementary therapy, may help to reduce inconvenience caused by the disease, treatments and their side effects (asthenia, anxiety and pain).

The main objective is to assess the impact of osteopathic treatment on pain in patients following breast cancer surgery. The impact will be considered beneficial if the pain score (digital scale) in the intervention group is lower, by at least two points, than the pain score in the control group at the end of the study.

This is a monocentric, randomized, parallel group, single-blind and prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman
* Surgery for a malignant breast tumor with sentinel lymph node technique
* Patient affiliated to a social security system
* Willing and able to provide written informed consent

Exclusion Criteria:

* Under-age women
* Pregnant woman
* Surgery for a malignant breast tumor with lymph node dissection
* Receiving adjuvant therapy during the study
* Receiving physiotherapy sessions (other than those made in immediate post-operative)
* Participating in the space "Au Fil de Soi": relaxing body massage and Energy Resonance by Cutaneous Stimulation (RESC)
* Person under guardianship or supervision
* Patient with impaired cognitive functions or lack of understanding of the French language
* Presenting a contraindication for osteopathy (major infectious and inflammatory conditions, trauma and other severe diseases)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at Day 9
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at day 20
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at day 26
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at Day 34
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at Day 40
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).
Assess the impact of osteopathic treatment on pain in patients following breast cancer surgery | at Day 48
  The primary outcome measure will be the evaluation of the "usual pain in the last eight days" measured from the pain score (digital scale). The pain score consists of asking the patient to quantify her pain on a virtual scale from 0 (absent pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 9
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 20
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 26
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 34
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 40
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the quality of life in patients who have been operated on breast cancer. | at day 48
  Assessment of quality of life by the SF-12 questionnaire, which is a shortened version of the " Medical Outcomes Study Short-Form General Health Survey " (SF-36), comprising only 12 of the 36 issues. The SF-12 is used to calculate two scores, which measure the functional health and well-being of the patient.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 9
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 20
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 26
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 34
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 40
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.
Assess the impact of osteopathic treatment on the reduction of anxiety of patients operated for breast cancer. | at Day 48
  Assessment of anxiodepressive disorders from the HAD scale (Hospital and Anxiety Depression), each response is rated from 0-3 on a scale evaluating semi-quantitatively the intensity of symptoms during the past week. This study will use just the score of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gil DUBERNARD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de gynécologie, Lyon, France